CLINICAL TRIAL: NCT07363317
Title: Effectiveness of Social Media-Based Educational Intervention (WhatsApp) on Dental Health Knowledge, Practices, and Attitudes Among Primary School Children Aged 10-12 Years in Cairo, Egypt: A Quasi-Experimental Study
Brief Title: Assessing the Impact of a Social Media-Based Educational Intervention Using WhatsApp Video Messages on Dental Caries Prevention Knowledge, Oral Hygiene Practices, and Attitudes Toward Dental Health Among Primary School Children Aged 10-12 Years in Public Schools in Cairo Governorate, Egypt: A Quasi-
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rana Mohamed Ahmed Farghal (Other)
Collaborators: Military Medical Academy, Bulgaria (Other); Cairo University (Other)
Responsible Party: Sponsor-Investigator, Rana Mohamed Ahmed Farghal, Technical Advisor, Office of the Egyptian Minister of Health and Population, Military Medical Academy,Egypt
Organization: Military Medical Academy,Egypt (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MMA-DENT-2026-001
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Dental Caries; Oral Health Behavior Change; Oral Hygiene, Oral Health; Knowledge, Attitudes, Practice; Child Behavioral Health; Preventive Health Care
Keywords: Dental Health Education; WhatsApp; Mobile Health; Children Oral Health; Primary School Children; Dental Caries Prevention; Video-Based Learning; Oral Hygiene
MeSH Terms: conditions — Dental Caries; Behavior

STUDY DESIGN:
Intervention Model Description: This is a two-arm parallel group quasi-experimental study. Participants are assigned to one of two groups based on grade level at enrollment and remain in their assigned group throughout the 8-week study period. The intervention group (Grade 5 students, n=75) receives six educational videos about dental health delivered via WhatsApp over 6 weeks (one video per week). The control group (Grade 6 students, n=75) continues usual school and home activities without receiving study-related educational materials during the study period. Both groups are assessed at baseline (Week 0) and post-intervention (Week 8) using identical questionnaires measuring dental health knowledge, practices, and attitudes. This parallel design was chosen to minimize contamination between groups by utilizing different grade levels that have limited daily interaction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Grade 5 students (n=75) who receive six educational videos about dental health delivered via WhatsApp over 6 weeks (one video per week, posted every Monday at 4:00 PM). Videos are 2-5 minutes long and cover: Week 1 - Why teeth are important, Week 2 - Proper brushing technique, Week 3 - Foods that harm teeth, Week 4 - Foods good for teeth, Week 5 - Importance of dental visits, Week 6 - Fun tips for healthy smiles. All videos are in Arabic with colorful animations appropriate for children aged 10-12 years. Children are assessed at baseline (Week 0) and post-intervention (Week 8).
  Interventions: Behavioral: WhatsApp-Based Dental Health Education for Children
- Control Group (No Intervention): Grade 6 students (n=75) who continue their usual school curriculum and home activities without receiving study-related educational materials during the 8-week study period. Children are assessed at baseline (Week 0) and at Week 8 using the same questionnaires as the intervention group. After completing post-intervention assessments, this group will be invited to join a separate WhatsApp group to receive all six educational videos for ethical reciprocity.

INTERVENTIONS:
Behavioral: WhatsApp-Based Dental Health Education for Children — Six educational videos about dental health delivered via a closed WhatsApp group over 6 weeks (one video per week, posted every Monday at 4:00 PM). Each video is 2-5 minutes long, features Arabic voiceover with colorful animations, and is age-appropriate for children aged 10-12 years. Video topics: Week 1 - Importance of teeth (anatomy, functions, consequences of tooth loss), Week 2 - Proper brushing technique (circular motion, all surfaces, 2-minute duration, twice daily), Week 3 - Foods that harm teeth (sugary foods, sticky snacks, frequent eating), Week 4 - Foods good for teeth (calcium-rich foods, crunchy vegetables, water), Week 5 - Importance of dental visits (professional cleaning, preventive care, reducing fear), Week 6 - Fun tips for healthy smiles (review, establishing routines, positive reinforcement). All videos selected based on evidence-based content aligned with WHO and American Academy of Pediatric Dentistry guidelines.
  Other Names: Social Media-Based Oral Health Promotion; Digital Dental Health Education Program; mHealth Educational Intervention; Video-Enhanced Health Literacy Intervention
  Arms: Intervention Group

SUMMARY:
The goal of this study is to learn if educational videos sent through WhatsApp can improve dental health knowledge, healthy habits, and attitudes in primary school children aged 10 to 12 years in Cairo, Egypt.

The main questions it aims to answer are:

* Do children who receive dental health videos through WhatsApp have better knowledge about caring for their teeth after 8 weeks compared to children who do not receive the videos?
* Do children who watch the videos brush their teeth more often and correctly, and make healthier food choices?
* Do children who watch the videos feel more positive about taking care of their teeth and visiting the dentist?

Researchers will compare children in Grade 5 who receive 6 short dental health videos through WhatsApp (one video per week for 6 weeks) to children in Grade 6 who continue their normal school activities to see if the videos lead to better knowledge, healthy habits, and more positive attitudes about dental health.

Participants will:

* Answer questions about their dental health knowledge, tooth brushing and eating habits, and feelings about dental care at the start of the study (takes about 15 to 20 minutes in a private room at school)
* Children in Grade 5 will join a WhatsApp group and receive one short video (2 to 5 minutes) each week for 6 weeks about topics like why teeth are important, how to brush teeth correctly, which foods are goo

DETAILED DESCRIPTION:
STUDY DESIGN AND RATIONALE

This is a quasi-experimental pre-post study with a non-equivalent control group. The study compares WhatsApp-delivered video-based educational intervention (intervention group) to standard school activities (control group) among primary school children aged 10-12 years in Cairo, Egypt.

Quasi-experimental design was chosen because randomization at the individual level was not feasible in the school setting. To minimize contamination between groups, children were assigned by grade level: all Grade 5 students form the intervention group, and all Grade 6 students form the control group. This approach reduces daily interaction between groups while maintaining comparable baseline characteristics.

The intervention is based on social cognitive theory, which emphasizes observational learning, self-efficacy, and behavioral modeling. Videos were selected to demonstrate proper techniques, provide positive role models, and build confidence in children's ability to practice good oral health behaviors.

INTERVENTION DESCRIPTION

Intervention Group (Grade 5, n=75):

Children will receive 6 educational videos about dental health via a closed WhatsApp group over 6 weeks (one video per week, posted every Monday at 4:00 PM).

Video Content and Delivery Schedule:

Week 1 - "Why Do We Need Teeth?" (3:58 minutes) Topics: Dental anatomy and tooth functions (chewing, speaking, smiling), consequences of tooth loss, importance of caring for baby teeth, introduction to tooth decay. Format: Animated educational video with Arabic voiceover.

Week 2 - "The Right Way to Brush Our Teeth" (4:17 minutes) Topics: Step-by-step brushing technique (circular motion), brushing all surfaces (outer, inner, chewing), tongue brushing, frequency (twice daily), duration (2 minutes), replacing toothbrush every 3 months. Format: Animated demonstration with catchy song and visual instructions.

Week 3 - "Foods That Harm Our Teeth" (3-4 minutes) Topics: How sugary foods and drinks feed bacteria to produce acid causing cavities, sticky foods, frequent snacking, identifying unhealthy foods (candy, soda, cookies), limiting sugar intake. Format: Interactive animated video with visual categorization.

Week 4 - "Foods Good for Our Teeth" (3-4 minutes) Topics: Calcium-rich foods (milk, cheese, yogurt) strengthen teeth, crunchy fruits and vegetables naturally clean teeth, water rinses the mouth, importance of balanced diet for oral health. Format: Animated educational video.

Week 5 - "Why Do We Go to the Dentist?" (2-4 minutes) Topics: What happens during a dental checkup (examination, cleaning), professional cleaning removes plaque, importance of preventive care, recommended visit frequency (every 6 months), making dental visits fun instead of scary. Format: Animated story or live-action video showing positive dental visit experience.

Week 6 - "Fun Tips for Healthy Teeth" (2-3 minutes) Topics: Review of key messages, creative ways to make brushing fun (brushing to a song for 2 minutes, family brushing time, friendly competitions), establishing morning and evening routines, celebrating healthy smiles, positive reinforcement and encouragement. Format: Musical video with children singing and performing.

All videos were selected based on: high-quality production (clear audio/video), evidence-based content (aligned with WHO and American Academy of Pediatric Dentistry guidelines), age-appropriateness (10-12 years), cultural relevance (Arabic language, Egyptian context), engaging format (animation, demonstration, music), appropriate length (2-5 minutes), positive tone (encouraging, not fear-based), no commercial content, educational value, and positive viewer feedback.

WhatsApp Group Management:

A closed WhatsApp group named "Healthy Teeth Friends" will include 75 intervention group children and approximately 45 parents (60%) who optionally choose to join, with the researcher as group administrator.

Each weekly post includes: friendly greeting in Arabic, 2-3 sentence introduction about the week's topic, YouTube video link, encouraging message, and relevant emoji. Mid-week reminders will be sent to children who have not viewed the video within 48 hours. The researcher will monitor the group daily, respond to questions within 24 hours, and document intervention fidelity including date/time of posting, number of views within 48 hours, number of questions and reactions, and responses provided.

Control Group (Grade 6, n=75):

Children will continue their usual school and home activities without receiving study-related educational materials during the 8-week study period. They will be informed that a second assessment will occur in May. After completing post-intervention assessments, the control group will be invited to a separate WhatsApp group to receive all 6 educational videos for ethical reciprocity.

OUTCOME MEASURES

Primary Outcome:

Dental Health Knowledge

ELIGIBILITY:
Inclusion Criteria:

* Children aged 10 to 12 years (Grades 5 or 6)
* Enrolled in the selected public primary school in Cairo, Egypt
* Able to understand and speak Arabic
* Parent or legal guardian provides written informed consent
* Child provides verbal assent to participate
* Child or parent has access to a smartphone with WhatsApp (for intervention group only)
* Child or parent willing to join WhatsApp group and view educational videos (for intervention group only)
* Able to complete questionnaire interview in Arabic

Exclusion Criteria:

* Children with severe cognitive or developmental disabilities that would prevent understanding questionnaire items or educational content
* Children with serious chronic medical conditions requiring intensive medical care that would interfere with study participation
* Children who are unable to attend school regularly (more than 2 days absence per week on average)
* Children who plan to transfer to another school during the study period (8 weeks)
* Children whose parents refuse consent or who refuse to provide assent
* Children currently participating in another dental health education program or clinical trial
* For intervention group: children or parents without smartphone access or unwilling to use WhatsApp

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Dental Health Knowledge Score | Baseline (Week 0) and 8 weeks after baseline
  Change in dental health knowledge from baseline to Week 8, measured using a validated 10-item questionnaire. Each correct answer scores 1 point (total score range 0-10, with higher scores indicating better knowledge). Questions assess knowledge about tooth anatomy and functions, causes of tooth decay, proper brushing technique, recommended brushing frequency and duration, beneficial and harmful foods for teeth, and importance of regular dental visits. Good knowledge is defined as a score of 8 or higher out of 10. The primary outcome is the mean change in knowledge score between baseline and Week 8.

SECONDARY OUTCOMES:
Change in Dental Health Practices Score | Baseline (Week 0) and 8 weeks after baseline
  Change in oral health practices from baseline to Week 8, measured using a validated 9-item questionnaire (total score range 0-18, with higher scores indicating better practices). Items assess toothbrushing frequency (twice daily), duration (2 minutes), technique (all tooth surfaces), fluoride toothpaste use, consumption of sugary foods and drinks, eating between meals, eating sweets before bed, rinsing mouth after meals, and eating vegetables and fruits. Each item scores 0-2 points based on adherence to recommended practices. Good practices are defined as a score of 13 or higher out of 18. The outcome is the mean change in practices score between baseline and Week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Passant Nagi, PHD, Study Director — Cairo University, Military Medical Academy; Rana M FARGHAL, B.D.S., Principal Investigator — Military Medical Academy, Bulgaria
Locations (1):
- Mount International School, New Administrative Capital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect the privacy of child participants and comply with ethical approval conditions. Summary results will be publicly available through the study's published thesis, peer-reviewed journal articles, and aggregate results posted on ClinicalTrials.gov.

REFERENCES:
- [Background] Soldani F, Wu J. School based oral health education. Evid Based Dent. 2018 Jun;19(2):36-37. doi: 10.1038/sj.ebd.6401298. PMID 29930371
- [Result] Towle-Miller LM, Miecznikowski JC, Zhang F, Tritchler DL. SuMO-Fil: Supervised multi-omic filtering prior to performing network analysis. PLoS One. 2021 Aug 3;16(8):e0255579. doi: 10.1371/journal.pone.0255579. eCollection 2021. PMID 34343218
- [Result] Cooper AM, O'Malley LA, Elison SN, Armstrong R, Burnside G, Adair P, Dugdill L, Pine C. Primary school-based behavioural interventions for preventing caries. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD009378. doi: 10.1002/14651858.CD009378.pub2. PMID 23728691
- [Result] Social Media Interventions Chen Y, Smith M, Johnson K. Social media interventions for health promotion among adolescents and young adults: A meta-analysis. Digital Health. 2025;11:20552076251234568.
- [Result] Type: Other Full Citation: Hassan NM, Gaber A, El-Sayed MH. Oral health status, knowledge, and behaviors among school children in Cairo, Egypt, and their impact on quality of life. Clinical, Cosmetic and Investigational Dentistry. 2019;11:369-380.
- See also: WHO oral health guidelines and school health programs — https://www.who.int/health-topics/oral-health
- See also: Egyptian Ministry of Health and Population - School health initiatives — https://www.mohp.gov.eg